CLINICAL TRIAL: NCT00820885
Title: A Double-Blind Multi-Dose Tolerability and Pharmacokinetic Study of Teduglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: CL0600-022
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Pharmacokinetics and Safety of Elevated Doses
MeSH Terms: interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- cohort A (Other): 20 mg dose 20 mg/ML concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort AR (Other): 20 mg in 50 mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort C (Other): 25 mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort D (Other): 15 mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort E (Other): 10 mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort F (Other): 30mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- Cohort H (Other): 50mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide
- cohort I (Other): 80mg in 50mg/ml concentration and placebo
  Interventions: Drug: teduglutide; Drug: tedguglutide

INTERVENTIONS:
Drug: teduglutide — subcutaneous injection given once a day in the abdomen. Drug is lypholized powder.
  Other Names: Gattex is the brand name
Drug: teduglutide — Once daily subcutaneous injection in the abdomen. Drug is lypholized powder reconstituted with sterile water
  Other Names: Gattex
Drug: tedguglutide — lypholized powder reconstituted with sterile water and injection subcutaneously once a day in the abdomen.
  Other Names: Gattex

SUMMARY:
The primary objective of the study was to study the safety and tolerability of teduglutide following a once or possibly twice daily subcutaneous injection for eight consecutive days in healthy subjects. A secondary objective was to study the pharmacokinetics of teduglutide following a once or possibly twice daily injection for eight consecutive days in healthy subjects.

DETAILED DESCRIPTION:
Healthy subjects are enrolled once they have been screened and it is determined they qualify. The subjects are randomized to either placebo or the dose of teduglutide as outlined by the protocol at a 1:3 ratio. They will be injected with investigational product for eight consecutive days, with measurements taken including safety.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 55 years of age
* BMI of 18-35 inclusive
* Able to understand and sign informed consent form
* Willing and able to be confined at the clinical research center 8.5 days
* Women who are post-menopausal, surgically sterilized, or agree to use effective form of birth control
* Women of child bearing potential with a negative pregnancy test at screening and check-in
* Medically healthy with normal clinical results and ECG/lab profiles at screening and check-in

Exclusion Criteria

* Donated 1 pint or more of blood/blood products within 56 days prior to study or received plasma within 7 days prior to study
* Pregnancy or become pregnant
* Participated in another investigational trial 30 days prior
* Physical examination/medical history indicates clinical condition or concurrent illness unsuitable for study
* History/presence of clincally significant disease of any body system
* History/evidence of congenital hon-hemolytic hyperbilirubinemia
* History/evidence of gall stone disease, stomach or intestinal surgery
* History/evidence of colorectal cancer
* History/evidence of GI disease, e.g., malabsorption, Crohn's Disease, etc.
* History/evidence of skin rashes or dermatitis
* Taking prescription or over the counter medication (with the exception of oral contraception) during the 7 days preceding confinement to the clinical unit

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2006-09-06 (Actual); Primary Completion 2007-04-23 (Actual); Study Completion 2007-04-23 (Actual)

PRIMARY OUTCOMES:
Each dose arm is safe | Within 1 week of each cohort completion

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Northwest Kinetics, Tacoma, Washington, United States